CLINICAL TRIAL: NCT06466824
Title: Observational Study on the Outcome of Patients With Primary Immune Thrombocytopenia (ITP) Who Underwent Splenectomy After January 1st, 2010
Brief Title: Observational Study on the Outcome of Patients With ITP Who Underwent Splenectomy After 2010
Status: Not yet recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: ITP1324
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: splenectomy
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective data collection on ITP patients who underwent splenectomy from 01/01/2010 to 12/31/2022. The expected enrollment period is 6 months. The observation period of the enrolled patients is at least 1 year.

DETAILED DESCRIPTION:
Observational, longitudinal, retrospective study on ITP patients. Patients with ITP who underwent splenectomy from 01/01/2010 to 12/31/2022 will be enrolled. All useful data will be collected exclusively through consultation of outpatient medical records. The expected enrollment period is 6 months. The observation period of the enrolled patients is at least 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with primary ITP according to international criteria [2], who underwent to splenectomy from 01/01/2010 to 12/31/2022.
* Obtaining Informed Consent.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ITP who underwent splenectomy from 01/01/2010 to 12/31/2022 will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
evaluation of complications' incidence after splenectomy | at 90 days
  Determine the percentage and incidence of thrombotic, hemorrhagic and infectious complications occurring during the patient's follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Vianelli, Principal Investigator — UO Ematologia AOU Policlinico S.Orsola-Malpighi di Bologna